CLINICAL TRIAL: NCT00846326
Title: A Proof of Concept Study to Evaluate if Concomitant Topical Intranasal Steroid Prevents Tolerance and Rebound Congestion Due to Regular Oxymetazoline in Persistent Allergic Rhinitis.
Brief Title: Preventing Tolerance to Oxymetazoline in Allergic Rhinitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The suppliers were unable to provide the investigational medicinal product (IMP)
Sponsor: Brian J Lipworth (Other)
Responsible Party: Sponsor-Investigator, Brian J Lipworth, Professor (Clinical) Airway allergy and COPD, University of Dundee
Organization: University of Dundee (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VAI01
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Allergic Rhinitis; Tachyphylaxis; Rhinitis Medicamentosa
Keywords: allergic rhinitis; rhinitis medicamentosa; imidazolines; corticosteroid
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Oxymetazoline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxymetazoline-Fluticasone Propionate (Experimental): Combination nasal spray with oxymetazoline 0.05% and fluticasone propionate 0.05%
  Interventions: Drug: oxymetazoline-fluticasone propionate
- Oxymetazoline-placebo (Placebo Comparator): oxymetazoline 0.05% w/v and placebo fluticasone propionate
  Interventions: Drug: Oxymetazoline

INTERVENTIONS:
Drug: oxymetazoline-fluticasone propionate — Oxymetazoline 0.05% w/v Fluticasone propionate 0.05% w/w 2 squirts in each nostril twice daily
  Arms: Oxymetazoline-Fluticasone Propionate
Drug: Oxymetazoline — oxymetazoline 0.05% w/v and placebo nasal spray 2 squirts in each nostril twice daily
  Arms: Oxymetazoline-placebo

SUMMARY:
The investigators wish to evaluate the effects of decongestants like oxymetazoline and the lessening of this effect with time called 'tolerance'. The investigators will demonstrate a reversal of this tolerance with nasal steroids i.e. the investigators will show that nasal steroids protect against tolerance. This will tell us more on how the investigators can make this treatment effective and safe for patients suffering with allergic rhinitis.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) affects upto 25% of the worldwide population and is associated with asthma, with Scotland having the highest prevalence in the world. Nasal blockage is the main symptom of allergic rhinitis. Nasal blockage affects sleep quality and impairs daytime performance. It is a major cause of sickness absenteeism and has been shown to adversely affect quality of life. The most efficacious class of drugs for nasal blockage in AR are the nasal decongestants (sympathomimetics acting on alpha receptors which unblock the nose). These are available over the counter for routine use by people experiencing nasal blockage. Nasal steroids are the most effective drugs for overall symptoms of allergic rhinitis and are considered first line therapy by recent guidelines. There is widespread belief that prolonged use of decongestant sprays like oxymetazoline can result in a condition of decreased effectiveness called tolerance. It is thought that with time they lose their effectiveness and more and more medication is needed to achieve the same level of decongestion. Also it has been proposed that once stopped, the patient experiences rebound congestion. Long term users of nasal decongestants cannot get off their sprays because of this vicious cycle. These sprays act via stimulating the alpha adrenoreceptors in the nose. It is a poorly understood condition and the mechanism of action is unclear. What is also not clear is the time to onset of tolerance. From studies in the lung we know that tolerance in certain types of adrenoreceptors can be reversed by use of corticosteroids. We have also seen over many years of clinical practice that concomitant use of steroid sprays and decongestants prevents the onset of tolerance and rebound. Anecdotally, patients are often treated with this combination in clinic particularly during a common cold, hayfever season with high pollen counts and acute exacerbations. Therefore, we would like to conduct a proof of concept study to show that a combination nasal spray of decongestant and steroid protects against tolerance. We will also show protection against early rebound congestion. This will enable a new lease of life for allergic rhinitis sufferers, whose quality of life is most affected by nasal blockage and the absence of an effective long term drug strategy for it.

ELIGIBILITY:
Inclusion Criteria:

* Male of Female aged 18-65 years.
* Persistent allergic rhinitis with or without asthma.
* Atopy to atleast one allergen on SPT.
* PNIF < 120 L/min (best of 3) and reversibility with OXY >20L/min.
* Ability to give a written informed consent.
* Ability and willingness to comply with the requirements of the protocol.

Exclusion Criteria:

* Recent respiratory tract/sinus infection within the last 2 months. .
* Pregnancy, planned pregnancy or lactation.
* Known or suspected hypersensitivity to any of the IMP's.
* Concomitant use of medicines (prescribed, OTC or herbal) like alpha blockers that may interfere with the trial.
* Nasal Polyposis grade 2+, Deviated nasal septum ≥ 50%
* The use of oral corticosteroids within the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the difference in peak PNIF response to incremental doses of Oxymetazoline [i.e. as a dose response] | Pre dose response, after 25, 50, 100, 200 mg/ml of oxymetazoline nasal spray

SECONDARY OUTCOMES:
Active Anterior Rhinomanometry | Pre dose response, after 25, 50, 100, 200 mg/ml of oxymetazoline nasal spray
Laser Doppler Velocimetry for nasal blood flow | Pre dose response, after 50 mg/ml Oxymetazoline and after 200 mg/ml of Oxymetazoline
Overnight urinary cortisol creatinine ratio | post run-in,2 weeks, 4 weeks
Nasal nitric oxide levels | after run-in, 2 weeks, 4 weeks
Serum eosinophils, ECP | post run-in, 2 weeks, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lipworth, MD, FRCP, Principal Investigator — University of Dundee
Locations (2):
- United Kingdom (2):
  - Ninewells Hospital and Medical School (Tayside NHS Trust, University of Dundee), Dundee
  - Perth Royal Infirmary (Tayside NHS Trust), Perth

REFERENCES:
- [Background] Bousquet J, Van Cauwenberge P, Khaltaev N; Aria Workshop Group; World Health Organization. Allergic rhinitis and its impact on asthma. J Allergy Clin Immunol. 2001 Nov;108(5 Suppl):S147-334. doi: 10.1067/mai.2001.118891. No abstract available. PMID 11707753
- [Background] Nassef M, Shapiro G, Casale TB; Respiratory and Allergic Disease Foundation. Identifying and managing rhinitis and its subtypes: allergic and nonallergic components--a consensus report and materials from the Respiratory and Allergic Disease Foundation. Curr Med Res Opin. 2006 Dec;22(12):2541-8. doi: 10.1185/030079906x158057. PMID 17265594
- [Background] Nolte H, Nepper-Christensen S, Backer V. Unawareness and undertreatment of asthma and allergic rhinitis in a general population. Respir Med. 2006 Feb;100(2):354-62. doi: 10.1016/j.rmed.2005.05.012. Epub 2005 Jul 11. PMID 16005621
- [Background] Gupta R, Sheikh A, Strachan DP, Anderson HR. Burden of allergic disease in the UK: secondary analyses of national databases. Clin Exp Allergy. 2004 Apr;34(4):520-6. doi: 10.1111/j.1365-2222.2004.1935.x. PMID 15080802
- [Background] Ferguson BJ. Influences of allergic rhinitis on sleep. Otolaryngol Head Neck Surg. 2004 May;130(5):617-29. doi: 10.1016/j.otohns.2004.02.001. PMID 15138430
- [Background] Patou J, De Smedt H, van Cauwenberge P, Bachert C. Pathophysiology of nasal obstruction and meta-analysis of early and late effects of levocetirizine. Clin Exp Allergy. 2006 Aug;36(8):972-81. doi: 10.1111/j.1365-2222.2006.02544.x. PMID 16911353
- [Background] Graf P. Long-term use of oxy- and xylometazoline nasal sprays induces rebound swelling, tolerance, and nasal hyperreactivity. Rhinology. 1996 Mar;34(1):9-13. PMID 8739860
- [Background] Ramey JT, Bailen E, Lockey RF. Rhinitis medicamentosa. J Investig Allergol Clin Immunol. 2006;16(3):148-55. PMID 16784007
- [Background] Petruson B. Treatment with xylometazoline (Otrivin) nosedrops over a six-week period. Rhinology. 1981 Sep;19(3):167-72. PMID 6171024
- [Background] Yoo JK, Seikaly H, Calhoun KH. Extended use of topical nasal decongestants. Laryngoscope. 1997 Jan;107(1):40-3. doi: 10.1097/00005537-199701000-00010. PMID 9001263
- [Background] Watanabe H, Foo TH, Djazaeri B, Duncombe P, Mackay IS, Durham SR. Oxymetazoline nasal spray three times daily for four weeks in normal subjects is not associated with rebound congestion or tachyphylaxis. Rhinology. 2003 Sep;41(3):167-74. PMID 14579657
- [Background] Hallen H, Enerdal J, Graf P. Fluticasone propionate nasal spray is more effective and has a faster onset of action than placebo in treatment of rhinitis medicamentosa. Clin Exp Allergy. 1997 May;27(5):552-8. PMID 9179430
- [Background] Tan KS, Grove A, McLean A, Gnosspelius Y, Hall IP, Lipworth BJ. Systemic corticosteriod rapidly reverses bronchodilator subsensitivity induced by formoterol in asthmatic patients. Am J Respir Crit Care Med. 1997 Jul;156(1):28-35. doi: 10.1164/ajrccm.156.1.9610113. PMID 9230722
- [Background] Hamamdzic D, Duzic E, Sherlock JD, Lanier SM. Regulation of alpha 2-adrenergic receptor expression and signaling in pancreatic beta-cells. Am J Physiol. 1995 Jul;269(1 Pt 1):E162-71. doi: 10.1152/ajpendo.1995.269.1.E162. PMID 7631772
- [Background] Davies AO, Lefkowitz RJ. Regulation of beta-adrenergic receptors by steroid hormones. Annu Rev Physiol. 1984;46:119-30. doi: 10.1146/annurev.ph.46.030184.001003. No abstract available. PMID 6324653